CLINICAL TRIAL: NCT03000088
Title: Stylet Angle for McGrath Videolaryngoscopy
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Lee, Clinical assistant prefessor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-DE4-15-414
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Intubation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 60° angle group: intubate using McGrath Videolaryngoscope with 60° angled stylet
  Interventions: Device: intubate with 60° angled stylet
- 90°angle group: intubate using McGrath Videolaryngoscope with 90° angled stylet
  Interventions: Device: intubate with 60° angled stylet

INTERVENTIONS:
Device: intubate with 60° angled stylet
  Groups: 60° angle group
Device: intubate with 60° angled stylet
  Groups: 90°angle group

SUMMARY:
The McGrath videolaryngoscope (VL) provides excellent laryngoscopic views, but directing an endotracheal tube is not easy, so routine using of stylet is recommended. The goal of this study is to determine the appropriate angle of stylet by comparing time to intubation (TTI).

ELIGIBILITY:
Inclusion Criteria:

* an American Society of Anesthesiologists physical status (ASA) 1 or 2

Exclusion Criteria:

* a suspected difficult airway (Mallampati score Ⅳ)
* known cervical spine injury
* required rapid sequence induction
* emergency operation

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for elective surgery requiring orotracheal intubation in our hospital
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiyoung Lee, MD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients scheduled for elective surgery requiring orotracheal intubation in our hospital. The last patient completed in August 2016.
Groups:
- 60° Angle Group: intubate using McGrath Videolaryngoscope with 60° angled stylet
  intubate with 60° angled stylet
- 90°Angle Group: intubate using McGrath Videolaryngoscope with 90° angled stylet
  intubate with 60° angled stylet
Period: Overall Study
Arm/Group | 60° Angle Group | 90°Angle Group
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 60° Angle Group | 90°Angle Group | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (14) | 41 (14) | 41 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 54 | 57 | 111
Thyromental distance [Mean (Standard Deviation); unit: cm] | 9.2 (1.3) | 9.2 (1.4) | 9.2 (1.3)
Mouth opening [Median (Standard Deviation); unit: cm] | 5.4 (1.1) | 5.2 (0.9) | 5.3 (1.0)
range of motion of cervical spine [Count of Participants; unit: Participants]
  normal | 69 | 70 | 139
  reduced | 1 | 0 | 1
  fixed | 0 | 0 | 0
upper incisors status [Count of Participants; unit: Participants]
  normal | 68 | 70 | 138
  absent | 1 | 0 | 1
  fixed | 1 | 0 | 1
Mallampati score [Count of Participants; unit: Participants] — Lower Mallamlapti score predicts easier intubation than did higher Mallampati score.
  Participants
    Mallampati score 1 | 41 | 41 | 82
    Mallampati score 2 | 22 | 20 | 42
    Mallampati score 3 | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubation
Time Frame: 10 minutes around intubation
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 90°Angle Group | 60° Angle Group
Number analyzed (Participants) | 70 | 70
seconds | 32.5 (9.4) | 29.3 (6.4)

ADVERSE EVENTS:
Arm/Group | 60° Angle Group | 90°Angle Group
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No